CLINICAL TRIAL: NCT02332915
Title: Effect of Intensity of Treatment on Rehabilitation of Acquired Apraxia of Speech
Brief Title: Treatment Intensity - Apraxia of Speech
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C1782-R
Record Dates: First submitted 2014-12-22; First posted 2015-01-07 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-03

CONDITIONS: Aphasia; CVA; Apraxia of Speech
Keywords: apraxia; aphasia; rehabilitation; efficacy; intensity
MeSH Terms: conditions — Aphasia; Apraxias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPT - Intense First (Experimental): Participants will receive intense application in the first phase of treatment, followed by the non intense application of treatment.
  Interventions: Behavioral: Sound Production Treatment (SPT)
- SPT - Traditional First (Experimental): Participants will receive non intense, "traditional" application of treatment in the first phase of treatment, followed by the intense application of treatment.
  Interventions: Behavioral: Sound Production Treatment (SPT)

INTERVENTIONS:
Behavioral: Sound Production Treatment (SPT) — SPT is a behavioral treatment for acquired apraxia of speech. It involves verbal modeling of target words by the clinician, simultaneous productions, articulatory placement instructions, and repeated practice. Treatment is administered in the context of an hierarchy.

SUMMARY:
A growing neurorehabilitation literature suggests that intense treatment may be desired to maximize the effects of therapy following neurologic injury. This investigation is designed to facilitate the development of efficacious, clinically applicable treatment for acquired apraxia of speech by examining the effects of intensity of treatment (e.g., 9 hours per week vs. 3 hours per week, while holding total number of sessions constant) with a group of speakers who have chronic apraxia of speech and aphasia.

DETAILED DESCRIPTION:
This research was designed to examine the effects of treatment intensity on outcomes associated with an established treatment for acquired apraxia of speech (AOS). Intensity in the form of dose frequency and total intervention duration was evaluated with Sound Production Treatment (SPT). The investigators examined the effects of intense dose frequency (nine, one-hour sessions per week) and traditional dose frequency (three, one hour sessions per week). Total number of treatment sessions was held constant allowing for comparison of total intervention duration (27 sessions over 3 weeks versus 27 sessions over 9 weeks). A two-phase, group cross-over design was used. Thirty-six participants with chronic aphasia and AOS were recruited. Twenty-four participants completed then entire study and were quasi-randomly assigned to one of two treatment groups - intense first or traditional first (12 per group). One group received SPT applied with intense dose frequency (SPT-I) followed by SPT applied with traditional dose frequency (SPT-T). The other group received the treatments in the reverse order (SPT-T followed by SPT-I). A two week no treatment interval separated the treatment phases. The outcomes of interest addressed changes in trained and untrained speech behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Veterans and non Veterans
* Males or females
* Stroke survivor who is at least 4 months post-stroke
* Speaker of English since childhood
* Ability to pass a pure-tone hearing screening (aided or unaided)
* currently non-hospitalized
* Age 21 to 90 years

Exclusion Criteria:

* neurological condition other than stroke
* currently clinically depressed
* history of speech/language problems prior to stroke
* untreated psychopathology

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie L Wambaugh, PhD, Principal Investigator — VA Salt Lake City Health Care System, Salt Lake City, UT
Locations (2):
- United States (2):
  - VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania
  - VA Salt Lake City Health Care System, Salt Lake City, UT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
All of the following will be shared for de-identified participants: Individual participant experimental stimuli will be provided in publications. Individual participant probe performance data will be shared in publications. Individual effect size data will be shared in publications. Individual pretreatment assessment performance will be shared in publications.
Supporting Information: Study Protocol, SAP
Time Frame: Individual data for 17 participants has been shared in publications. The data for the remaining 7 participants will be shared in a final publication - approximately by January 2022.
Access Criteria: Individual data are available in publications.

REFERENCES:
- [Result] Wambaugh JL, Wright S, Boss E, Mauszycki SC, DeLong C, Hula W, Doyle PJ. Effects of Treatment Intensity on Outcomes in Acquired Apraxia of Speech. Am J Speech Lang Pathol. 2018 Mar 1;27(1S):306-322. doi: 10.1044/2017_AJSLP-16-0188. PMID 29497746
- [Result] Wambaugh JL, Wright S, Nessler C, Mauszycki SC, Bunker L, Boss E, Zhang Y, Hula WD, Doyle PJ. Further Study of the Effects of Treatment Intensity on Outcomes of Sound Production Treatment for Acquired Apraxia of Speech: Does Dose Frequency Matter? Am J Speech Lang Pathol. 2020 Feb 7;29(1):263-285. doi: 10.1044/2019_AJSLP-19-00005. Epub 2020 Feb 3. PMID 32011909

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SPT - Intense First | SPT - Traditional First
Started | 18 | 18
Completed | 12 | 12
Not Completed | 6 | 6
Not completed — Moved out of region | 3 | 0
Not completed — Unrelated illness | 1 | 1
Not completed — Travel distance prohibitive | 0 | 1
Not completed — did not meet inclusion criteria | 2 | 4

BASELINE CHARACTERISTICS:
Population: Persons with aphasia and apraxia of speech who completed both phases of treatment.
Groups:
- SPT - Intense First: Participants received intense application in the first phase of treatment, followed by the non intense application of treatment.
  Sound Production Treatment (SPT): SPT is a behavioral treatment for acquired apraxia of speech. It involves verbal modeling of target words by the clinician, simultaneous productions, articulatory placement instructions, and repeated practice. Treatment is administered in the context of an hierarchy.
  Intense application = SPT-I: treatment administered for 3 hourly sessions per day, 3 days per week, for 3 weeks for a total of 27 hourly sessions.
- SPT - Traditional First: Participants received non intense, "traditional" application of treatment in the first phase of treatment, followed by the intense application of treatment.
  Sound Production Treatment (SPT): SPT is a behavioral treatment for acquired apraxia of speech. It involves verbal modeling of target words by the clinician, simultaneous productions, articulatory placement instructions, and repeated practice. Treatment is administered in the context of an hierarchy.
  Traditional application = SPT-T: treatment administered for 1 hourly session, 3 days per week for 9 weeks for a total of 27 hourly sessions.
- Total: Total of all reporting groups
Arm/Group | SPT - Intense First | SPT - Traditional First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of participants in years
  years | 55.75 (13.07) | 61.83 (12.13) | 58.79 (12.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 12 | 11 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Accuracy of Articulation of Treated Items in Baseline (Pre-treatment) [Mean (Standard Deviation); unit: units on a scale] — Accuracy of articulation of items designated for treatment. Experimental words were produced in pre-treatment probes. Participant productions were scored as being correctly produced according to phonetic transcription. The baseline measure represents the percentage of words produced correctly on a scale ranging from 0% accuracy to 100% accuracy.
  units on a scale | 12.03 (6.14) | 10.5 (8.3) | 11.28 (7.19)
Accuracy of Articulation of UNtreated Items in Baseline (Pre-treatment) [Mean (Standard Deviation); unit: units on a scale] — Accuracy of articulation of items designated to not receive treatment; these items were phonetically similar to treated items. Experimental words were produced in pre-treatment probes. Participant productions were scored as being correctly produced according to phonetic transcription. The baseline measure represents the percentage of words produced correctly on a scale ranging from 0% accuracy to 100% accuracy.
  units on a scale | 14.07 (6.67) | 13.9 (9.98) | 13.99 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Articulation of TREATED ITEMS Measured as Effect Size - Change From Baseline to End of Treatment Phase
Description: Accuracy of articulation of sounds in words, phrases, sentences designated for treatment. Assessed in nontreatment probes with productions elicited through repetition. Change in accuracy of articulation of trained items was measured from baseline to 2 weeks post treatment using effect size calculations as the indicator of magnitude of change. Percent accuracy was calculated for each probe (maximum = 100%, minimum = 0% correct). Effect size calculations involved calculating the difference between post- and pre-treatment probe accuracy percentages with corrections made for variability (standard deviations in performance). The larger the effect size, the greater the change in performance from pre-treatment. Positive effect sizes = increases in accuracy & negative effect sizes = decreases in accuracy.
Time Frame: Pre treatment, 2 weeks following the first treatment phase, 2 weeks following the second treatment phase
Measure: Mean (Standard Deviation); unit: effect sizes; magnitude of change
Groups:
- SPT - Intense: All Participants: All participants received Sound Production Treatment (SPT). Half the participants received SPT applied in an intense manner (SPT-Intense; SPT-I) first for 27 sessions. Following a 2 week washout period, those participants then received SPT applied in non-intense fashion (SPT-Traditional; SPT-T) for 27 sessions. The other half of the participants received the treatments in the opposite order. All 24 administrations of SPT-Intense were analyzed relative to all 24 administrations of SPT-Traditional.
  Sound Production Treatment (SPT): SPT is a behavioral treatment for acquired apraxia of speech. It involves verbal modeling of target words by the clinician, simultaneous productions, articulatory placement instructions, and repeated practice. Treatment is administered in the context of an hierarchy.
- SPT - Traditional (Non-intense): All Participants: All participants received Sound Production Treatment (SPT). Half the participants received SPT applied in a non-intense manner (SPT- Traditional; SPT-T) first for 27 sessions. Following a 2 week washout period, those participants then received SPT applied in an intense fashion (SPT-Intense; SPT-I) for 27 sessions. The other half of the participants received the treatments in the opposite order. All 24 administrations of SPT-Intense were analyzed relative to all 24 administrations of SPT-Traditional.
  Sound Production Treatment (SPT): SPT is a behavioral treatment for acquired apraxia of speech. It involves verbal modeling of target words by the clinician, simultaneous productions, articulatory placement instructions, and repeated practice. Treatment is administered in the context of an hierarchy.
Arm/Group | SPT - Intense: All Participants | SPT - Traditional (Non-intense): All Participants
Number analyzed (Participants) | 24 | 24
effect sizes; magnitude of change | 19.7 (12.6) | 28.9 (17.2)
Statistical Analysis 1: Comparison: SPT - Intense: All Participants vs SPT - Traditional (Non-intense): All Participants; Null hypothesis is that there is no difference in mean effect size values for 2-week follow-up values for treated items for SPT-Intense and SPT-Traditional. The test was performed with a significance level of 0.05 (two-sided); Test type: Superiority; p = .0128, t-test, 2 sided; dependent t-test

2. Primary Outcome: Accuracy of Articulation of Untreated Items (Generalization) Measured as Effect Size - Change From Baseline to End of Treatment Phase
Description: Change in accuracy of articulation of untrained items as measured by effect sizes reflecting magnitude of change. Production of words designated to not receive treatment (i.e., generalization items) was measured repeatedly in non treatment probes prior to treatment, throughout all study phases, and at 2 weeks post treatment with percent accuracy calculated for each probe (0% to 100% correct). Effect size calculations involved calculating the difference between post- and pre-treatment probe accuracy percentages with corrections made for variability (standard deviations in performance). The larger the effect size, the greater the change in performance from pre-treatment.
Time Frame: Pre treatment, 2 weeks following the first treatment phase, 2 weeks following the second treatment phase
Population: 24 effect sizes from all 24 participants
Measure: Mean (Standard Deviation); unit: effect sizes; magnitude of change
Groups:
- SPT - Intense; All Participants: All participants received Sound Production Treatment (SPT). Half the participants received SPT applied in an intense manner (SPT-Intense; SPT-I) first for 27 sessions. Following a 2 week washout period, those participants then received SPT applied in non-intense fashion (SPT-Traditional; SPT-T) for 27 sessions. The other half of the participants received the treatments in the opposite order. All 24 administrations of SPT-Intense were analyzed relative to all 24 administrations of SPT-Traditional.
  Sound Production Treatment (SPT): SPT is a behavioral treatment for acquired apraxia of speech. It involves verbal modeling of target words by the clinician, simultaneous productions, articulatory placement instructions, and repeated practice. Treatment is administered in the context of an hierarchy.
- SPT - Traditional; All Participants: All participants received Sound Production Treatment (SPT). Half the participants received SPT applied in a non-intense manner (SPT- Traditional; SPT-T) first for 27 sessions. Following a 2 week washout period, those participants then received SPT applied in an intense fashion (SPT- Intense; SPT- I) for 27 sessions. The other half of the participants received the treatments in the opposite order. All 24 administrations of SPT-Intense were analyzed relative to all 24 administrations of SPT-Traditional.
  Sound Production Treatment (SPT): SPT is a behavioral treatment for acquired apraxia of speech. It involves verbal modeling of target words by the clinician, simultaneous productions, articulatory placement instructions, and repeated practice. Treatment is administered in the context of an hierarchy.
Arm/Group | SPT - Intense; All Participants | SPT - Traditional; All Participants
Number analyzed (Participants) | 24 | 24
effect sizes; magnitude of change | 7.9 (5.6) | 8.1 (8.9)
Statistical Analysis 1: Comparison: SPT - Intense; All Participants vs SPT - Traditional; All Participants; Null hypothesis is that there is no difference in mean effect size values for 2-week follow-up values for untreated (generalization) items for SPT-Intense and SPT-Traditional. The test was performed with a significance level of 0.05 (two-sided); Test type: Superiority; p = .942, t-test, 2 sided; dependent t-test

3. Secondary Outcome: Speech Intelligibility - Percent Intelligible Words Comparing Baseline to End of Treatment Phases
Description: Measure of how well an unfamiliar listener can understand speech. The Assessment of Intelligibility of Dysarthric Speech will be employed. The participant will repeat words which will be audiorecorded. A trained, but unfamiliar listener will orthographically transcribe the words that are produced. The transcriptions will be compared to the list of target (intended words) to determine a percentage of words that are correctly understood. The score may range from 0% to 100% of words understood.
Time Frame: Pre treatment & 2 weeks following each treatment phase
Population: Intense SPT First Arm: one participant's data was lost due to data storage problems & three participants moved out of the region after the first treatment phase; Non-intense SPT First Arm: one participant's data was lost due to data storage problems & one participant moved out of the region after the first treatment phase
Measure: Mean (Standard Deviation); unit: % Intelligible words
Groups:
- Intense SPT First: Participants who received SPT Intense first, followed by a 2 week washout period and then received SPT-non-intense (SPT Traditional)
- Non-Intense (Traditional) SPT First: Participants who received non-intense SPT first, followed by a two week washout period, and then received intense SPT
- Both Arms Combined: Intense First + Traditional First: All participants who received both treatment phases regardless of treatment order
Arm/Group | Intense SPT First | Non-Intense (Traditional) SPT First | Both Arms Combined: Intense First + Traditional First
Number analyzed (Participants) | 15 | 13 | 22
% Intelligible words
  Baseline % Intelligibility | 45.15 (33.9) | 46.15 (29.5) | 48.96 (31.92)
  2 weeks Post Treatment #1: % Intelligibility: number analyzed (Participants) | 14 | 12 | 22
  2 weeks Post Treatment #1: % Intelligibility | 54.3 (37.2) | 61.5 (30.5) | 60.5 (33.1)
  2 weeks Post Treatment #2: % Intelligibility: number analyzed (Participants) | 11 | 11 | 22
  2 weeks Post Treatment #2: % Intelligibility | 61.3 (34.9) | 68.7 (30.5) | 65 (32.2)
Statistical Analysis 1: Comparison: Both Arms Combined: Intense First + Traditional First; Null Hypothesis: No difference in pre-treatment and post-treatment intelligibility scores; Test type: Other; p < .001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Entire course of study which was approximately 26 weeks per participant: pretreatment/baseline period = 4 weeks + 3 weeks Treatment 1 + 2 weeks washout + 9 weeks Treatment 2 + follow-up at 2 and 8 weeks.
Description: All participants received two applications of SPT: intense application and non-intense (Traditional) application. Participants were grouped together for analyses by treatment type; this was due to the fact that all participants received both treatments and were observed in the same way for both treatments regardless of which treatment was received first. There were not adverse events and consequently, no need to examine adverse events by arm.
Arm/Group | SPT - Intense: All Participants | SPT - Traditional (Non-intense): All Participants
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT02332915/Prot_001.pdf
  • Statistical Analysis Plan (2020-10-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT02332915/SAP_000.pdf